CLINICAL TRIAL: NCT04762953
Title: Phase II Trial of Sequential Systemic Therapy Plus Intraperitoneal Paclitaxel in Gastric/GEJ Cancer Peritoneal Carcinomatosis (STOPGAP)
Brief Title: Study of Sequential Systemic Therapy + Intraperitoneal Paclitaxel in Gastric/GEJ Peritoneal Carcinomatosis
Acronym: STOPGAP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Maheswari Senthil, MD, Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20206178; UCI 20-87 (Other: UCI CFCCC)
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric Cancer; Peritoneal Carcinomatosis; Gastroesophageal Junction (GEJ) Adenocarinoma; Paclitaxel; 5-FU; Fluorouracil; Leucovorin
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Paclitaxel; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: This clinical trial is a non-randomized, open label, single arm clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SingleArm: Systemic therapy and IP Paclitaxel in Gastric/GEJ Cancer Peritoneal Carcinomatosis (Experimental): Patients will receive sequential intraperitoneal paclitaxel along with intravenous paclitaxel, 5-FU, and leucovorin on Days 1 and 8 of every 21 day cycle for 3 months.
  Interventions: Drug: Paclitaxel; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Paclitaxel — Intraperitoneal Paclitaxel
Drug: Paclitaxel — IV Paclitaxel
Drug: Leucovorin — IV Leucovorin
Drug: Fluorouracil — IV 5-FU
  Other Names: 5-FU

SUMMARY:
This is a phase II clinical trial assessing the safety and efficacy of sequential systemic and intraperitoneal (IP) chemotherapy in patients with primary gastric/gastroesophageal junction cancer with cytology positive peritoneal lavage and/or peritoneal carcinomatosis.

DETAILED DESCRIPTION:
Patients with histologically proven primary gastric or gastroesophageal junction (Siewert 3) adenocarcinoma with positive peritoneal cytology or peritoneal carcinomatosis detected by laparoscopy, laparotomy or imaging and without evidence of distant organ metastasis will be eligible for this study. Patients will undergo systemic therapy for 3-4 months at the discretion of the medical oncologist based on molecular makers (PD-L1, HER -2 neu, MSI). Patients without distant organ metastatic progression after completion of systemic chemotherapy, will undergo diagnostic laparoscopy and IP port placement. IP regimen will consist of IV Paclitaxel, 5- FU and Leucovorin and IP Paclitaxel. Paclitaxel 40 mg/m2 will be instilled into the peritoneal cavity through the IP port on days 1 and 8, repeated every 21 days for 3 months (3-4 cycles). Restaging imaging with CT and /or diffusion weighted MRI with contrast will be obtained 4-6 weeks after completion of IP chemotherapy. Based on response and extent of disease, patients will be triaged to one of the following treatment plans: stable disease or response and PCI >10 - continue IP chemotherapy regimen, progression - switch to second line regimen, response with PCI ≤ 10 and complete cytoreduction is feasible - consider cytoreduction surgery (CRS) with intraperitoneal chemotherapy (IPEC).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed primary gastric or gastroesophageal adenocarcinoma and have received a minimum of three months of first line systemic treatment without visceral metastatic progression
* Must have peritoneal cytology positive disease or peritoneal carcinomatosis detected by imaging, laparoscopy or laparotomy
* Age ≥ 18 -75 years
* Performance status: ECOG performance status ≤ 2 (Appendix A) . ECOG 2 allowed is attributed to malignancy (rather than comorbidities)
* Life expectancy of greater than 6 months
* Adequate organ and marrow function as defined below:

  1. Leukocytes: ≥ 2,000/mcL
  2. Absolute Neutrophil Count: ≥ 1,500/mcL
  3. Platelets: ≥ 80,000/mcL
  4. Total Bilirubin: within normal institutional limits
  5. AST(SGOT)/ALT(SPGT): ≤5 X institutional upper limit of normal
  6. Creatinine: < 1.5 X institutional upper limit of normal
  7. Hemoglobin: > 8.0 g/dL (may be transfused)
  8. Serum albumin: ≥ g/dL
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Systemic treatment for unresectable or metastatic disease for more than three months prior to enrollment
* Any evidence of distant, solid organ metastases (visceral (liver, lung, brain), bone, extra-abdominal)
* Any evidence of extensive retroperitoneal lymph node metastases not amenable to resection during gastrectomy
* Any evidence of small or large bowel obstruction with the exception of gastric outlet obstruction due to primary malignancy
* Uncontrolled intercurrent illness including, but not limited to, the following conditions:

  1. Ongoing or active infection
  2. Symptomatic congestive heart failure
  3. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event,) within 3 months before initiation of treatment
  4. Unstable angina pectoris
  5. Cardiac arrhythmia
* History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in-situ and not treated with systemic therapy.
* Inability to comply with study and follow-up procedures as judged by the Investigator
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Has an active infection requiring systemic therapy.
* Prior surgery that would preclude safe diagnostic laparoscopy and port placement
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participants with Progression Free Survival at 1-Year | 1 year
  Progression-free survival is defined as the duration of time from start of systemic treatment to time of progression, death, or clinical deterioration attributed to disease progression as judged by the investigator. Radiographic progression is defined using the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) as a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm and/or appearance of new lesions.
Incidence of Treatment-Emergent Adverse Events [Safety] | From date of study treatment initiation to first date of disease progression, toxicity, delay of treatment, or withdrawal of treatment, assessed up to 12 months after the last patient is enrolled.
  To evaluate the safety of IP paclitaxel and IV paclitaxel, 5-FU, and leucovorin in patients with primary gastric/GEJ adenocarinoma with peritoneal carcinomatosis determined by the incidence of treatment-emergent adverse events. Adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.

SECONDARY OUTCOMES:
Overall Survival of Participants | From initiation of systemic treatment to up to 12 months after last patient is enrolled or until death from any cause.
  To assess the overall survival of participants from the start of systemic treatment to the death from any cause.
Patient Reported Quality of Life Outcomes | From initiation of study treatment until patient is off study, assessed up to 12 months after the last patient has started treatment.
  To assess the quality of life of participants such as mobility, self-care, daily activities, pain/discomfort and anxiety/depression and a visual analog scale (VAS). VAS consists of endpoints labeled best imaginable health status at the top and worse imaginable health state at the bottom having numeric values of 100 and 0 respectively.

OTHER OUTCOMES:
Expression of Plasma and Ascites Exosomal Gene Signature (EXOSIG) | From date of registration to up to 12 months after last patient is enrolled.
  To assess the expression of plasma and ascites exosomal gene signature (EXO SIG) in patients with gastric cancer peritoneal carcinomatosis compared to healthy controls.
Correlation of Plasma and Ascite Exosomal Gene Signature (EXOSIG) to Treatment Response | From date of registration to up to 12 months after last patient is enrolled.
  To assess the correlation of changes in exosomal gene signature to treatment response in patients with gastric cancer peritoneal carcinomatosis.

CONTACTS AND LOCATIONS:
Overall Officials: Maheswari Senthil, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

REFERENCES:
- [Derived] Senthil M, Dayyani F. Phase II clinical trial of sequential treatment with systemic chemotherapy and intraperitoneal paclitaxel for gastric and gastroesophageal junction peritoneal carcinomatosis - STOPGAP trial. BMC Cancer. 2023 Mar 4;23(1):209. doi: 10.1186/s12885-023-10680-1. PMID 36870941